CLINICAL TRIAL: NCT00037076
Title: Hepatitis C Prevalence in Perinatally Infected HIV-Positive Children Enrolled in PACTG 219C
Brief Title: Prevalence of Hepatitis C Virus Infection in HIV-Infected Children
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PACTG P1028S; 11657 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2002-05-14; First posted 2002-05-15 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections; Hepatitis C
Keywords: HIV Seropositivity; Hepatitis C; Polymerase Chain Reaction; RNA, Viral; Prevalence; Disease Transmission, Vertical; Hepacivirus; Enzyme Immunoassay; GB virus C
MeSH Terms: conditions — HIV Infections; Hepatitis C; HIV Seropositivity

SUMMARY:
The purpose of this study is to find out how many children who are infected with HIV are also infected with hepatitis C virus (HCV).

HCV infection is a major health concern. HIV-infected adults who are co-infected with HCV appear to have more rapid HIV disease progression. There is little data on how widespread HCV is among children who are HIV-infected. Information from this study will help determine the need for future HCV studies. This study also will obtain blood samples for future testing for other hepatitis viruses such as hepatitis G virus (HGV or GB virus C).

DETAILED DESCRIPTION:
HCV infection is a major public health concern with worldwide seroprevalence estimated at 1 percent. HIV-infected adults co-infected with HCV appear to have accelerated HIV disease progression. There is little data on HCV prevalence in the pediatric HIV-infected population. This substudy will provide estimates of HCV prevalence among HIV-infected children and determine the need for future HCV natural history and treatment protocols. In addition, this substudy will archive samples from patients for future testing for other hepatitis viruses such as hepatitis G virus (HGV or GB virus C).

Patients participating in PACTG 219C are selected randomly to enroll into PACTG P1028S. Patients who agree to participate have a single blood draw for HCV antibody (Enzyme Immunoassay-EIA) testing and HCV RNA (Polymerase Chain Reaction-PCR) testing. An additional blood draw is necessary in the case of discordant results between the HCV EIA and HCV PCR. HCV-negative patients have 1 study visit. Patients with positive HCV test results have 2 visits. Patients with discordant HCV test results have 2 or 3 visits.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this substudy if they:

* Are between 1 year and 20 years of age.
* Were infected with HIV from the mother at or around the time of birth.
* Are enrolled in PACTG 219C.
* Children known to be HCV-infected will be permitted to enter the substudy.

Exclusion Criteria

Patients may not be eligible for this substudy if they:

* Have hemophilia.
* Contracted HIV through a route other than from the mother around the time of birth.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600
Dates: Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Schuval, Study Chair
Locations (39):
- United States (37):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Phoenix Childrens Hosp, Phoenix, Arizona
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - Univ of California, San Diego, San Diego, California
  - UCSF, Moffitt Hospital (Pediatric), San Francisco, California
  - Children's Hosp of Denver, Denver, Colorado
  - Connecticut Childrens Med Ctr (Pediatric), Farmington, Connecticut
  - Yale Univ Med School, New Haven, Connecticut
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Miami (Pediatric), Miami, Florida
  - Med College of Georgia, Augusta, Georgia
  - The Med Ctr Inc, Columbus, Georgia
  - Mt Sinai Hosp Med Ctr / Dept of Pediatrics, Chicago, Illinois
  - The Univ of Chicago Children's Hosp, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Children's Hospital at SUNY Downstate, Brooklyn, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Univ of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University (Pediatric), Durham, North Carolina
  - Childrens Hosp of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hosp for Children, Philadelphia, Philadelphia, Pennsylvania
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
- Puerto Rico (2):
  - Univ. of Puerto Rico, U. Children's Hospital AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Tajiri H, Miyoshi Y, Funada S, Etani Y, Abe J, Onodera T, Goto M, Funato M, Ida S, Noda C, Nakayama M, Okada S. Prospective study of mother-to-infant transmission of hepatitis C virus. Pediatr Infect Dis J. 2001 Jan;20(1):10-4. doi: 10.1097/00006454-200101000-00003. PMID 11176560
- [Background] Tillmann HL, Heiken H, Knapik-Botor A, Heringlake S, Ockenga J, Wilber JC, Goergen B, Detmer J, McMorrow M, Stoll M, Schmidt RE, Manns MP. Infection with GB virus C and reduced mortality among HIV-infected patients. N Engl J Med. 2001 Sep 6;345(10):715-24. doi: 10.1056/NEJMoa010398. PMID 11547740
- [Background] Xiang J, Wunschmann S, Diekema DJ, Klinzman D, Patrick KD, George SL, Stapleton JT. Effect of coinfection with GB virus C on survival among patients with HIV infection. N Engl J Med. 2001 Sep 6;345(10):707-14. doi: 10.1056/NEJMoa003364. PMID 11547739
- [Background] Thomas SL, Newell ML, Peckham CS, Ades AE, Hall AJ. A review of hepatitis C virus (HCV) vertical transmission: risks of transmission to infants born to mothers with and without HCV viraemia or human immunodeficiency virus infection. Int J Epidemiol. 1998 Feb;27(1):108-17. doi: 10.1093/ije/27.1.108. PMID 9563703
- [Background] Papaevangelou V, Pollack H, Rochford G, Kokka R, Hou Z, Chernoff D, Hanna B, Krasinski K, Borkowsky W. Increased transmission of vertical hepatitis C virus (HCV) infection to human immunodeficiency virus (HIV)-infected infants of HIV- and HCV-coinfected women. J Infect Dis. 1998 Oct;178(4):1047-52. doi: 10.1086/515668. PMID 9806033